CLINICAL TRIAL: NCT05536089
Title: ctDNA Methylation Used to Monitor Postoperative Relapse and Evaluate Adjuvant Chemotherapy Efficacy in Resected Stage I and Stage II (Without High Risk) Colorectal Cancer After Radical Resection
Brief Title: ctDNA Methylation Application in Postoperative Relapse and Adjuvant Chemotherapy Efficacy Evaluation
Status: Recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Recovery-C
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cancer Colorectal
Keywords: early detection
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ctDNA positive: Postoperative ctDNA positive
  Interventions: Diagnostic Test: a multi-locus blood-based assay
- ctDNA negative: Postoperative ctDNA negative
  Interventions: Diagnostic Test: a multi-locus blood-based assay

INTERVENTIONS:
Diagnostic Test: a multi-locus blood-based assay — Colorectal tumor-specific plasma ctDNA methylation markers detection

SUMMARY:
In this study, the investigators aimed to apply their previously developed multi-locus blood-based assay targeting circulating tumor DNA methylation to monitor postoperative relapse and evaluate adjuvant chemotherapy efficacy in resected stage I and stage II (without high risk) colorectal cancer after radical resection.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational, real-world study. Research objects: patients with surgically resectable colorectal cancer and ctDNA positive before surgery in stage I and stage II (without high risk). After giving fully informed consent, the participants will undergo the regular treatment according to NCCN guidelines. Serial analysis of ctDNA will be performed at specific time points including pre-treatment, postoperative week 3, postoperative 5 years ( every 3 months for the first 2 years, and every 6 months for the rest 3 years). Participants will be observed and examined during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed stage I/II (without high risk) colorectal cancer.
* Male or female ≥ 18 years of age on the day of signing informed consent.
* Patients need to receive surgical resection, and with ctDNA positive prior to resection of colorectal cancer (CRC).
* Patients must have a performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

* Personal history of colorectal cancer, colorectal adenoma or aerodigestive tract cancer.
* Induction of neoadjuvant systemic therapy prior to resection of CRC.
* Patient is pregnant or lactating.
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.
* Inadequate tumor material (either quality and quantity) to support circulating tumor DNA (ctDNA) analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to enrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
5y DFS | 5 years
  The 5-year disease free survival rate of the patients from both cohorts.
ctDNA methylation markers versus CT/MRI | 5 years
  ctDNA methylation predictors of outcome will be compared to CT/MRI

SECONDARY OUTCOMES:
3y DFS | 3 years
  The 3-year disease free survival rate of the patients from both cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: KeFeng Ding, Ph.D, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University; Rui Liu, Ph.D, Principal Investigator — Singlera Genomics Inc.
Locations (1):
- Second Affiliated Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cai G, Cai M, Feng Z, Liu R, Liang L, Zhou P; ColonAiQ Group; Zhu B, Mo S, Wang H, Lan X, Cai S, Xu Y, Wang R, Dai W, Han L, Xiang W, Wang B, Guo W, Zhang L, Zhou C, Luo B, Li Y, Nie Y, Ma C, Su Z. A Multilocus Blood-Based Assay Targeting Circulating Tumor DNA Methylation Enables Early Detection and Early Relapse Prediction of Colorectal Cancer. Gastroenterology. 2021 Dec;161(6):2053-2056.e2. doi: 10.1053/j.gastro.2021.08.054. Epub 2021 Sep 4. No abstract available. PMID 34487783